CLINICAL TRIAL: NCT03774706
Title: Role of Sublingual Misoprostol With or Without Intravenous Tranexamic Acid for Reducing Post-partum Hemorrhage During and After Hemorrhagic Cesarean Section: A Double-Blind Randomized Clinical Trial
Brief Title: Sublingual Misoprostol With or Without Intravenous Tranexamic Acid During Hemorrhagic Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/184/18
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; tranexamic acid; misoprostol
MeSH Terms: interventions — Misoprostol; Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: double-blind placebo randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be appropriately blinded; the participants, outcome assessors and the surgeon performing the procedure will be blinded to the medication type, which will be used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol with TA (Active Comparator): two tablets sublingual misoprostol plus IgM tranexamic acid in 100 ml saline by slow iv
  Interventions: Drug: Misoprostol; Drug: Tranexamic Acid
- Misoprostol with placebo to TA (Active Comparator): two tablets sublingual misoprostol plus placebo to tranexamic acid ( 110 ml saline) by slow iv
  Interventions: Drug: Misoprostol; Drug: placebo to tranexamic acid

INTERVENTIONS:
Drug: Misoprostol — two tablets misoprostol 400 μg sublingual
  Other Names: Active Comparator
Drug: Tranexamic Acid — two ampoules of tranexamic acid (1gm in 10 ml) in 100ml saline
  Other Names: active comparator
  Arms: Misoprostol with TA
Drug: placebo to tranexamic acid — placebo to tranexamic acid (110 ml saline)
  Other Names: Placebo
  Arms: Misoprostol with placebo to TA

SUMMARY:
Purpose to evaluates the effects of sublingual misoprostol with or without intravenous tranexamic acid (TA) on reducing post-partum hemorrhage during and after hemorrhagic cesarean section.

DETAILED DESCRIPTION:
Different uterotonic agents administration, mainly oxytocin, has been routinely used to reduce the frequency of cesarean section (CS) -related hemorrhage; however, some studies reported that oxytocin use in the setting of CS may result in maternal adverse effects, including hypotension and tachycardia., Therefore, investigating other therapeutic agents with lower adverse effects and higher efficacy is needed. Recently, a number of studies reported a correlation between fibrinogen decrease and cesarean-related hemorrhage. Furthermore, extensive tissue injury increases fibrinolysis by shifting the hemostatic equilibrium and contributing to bleeding. Therefore, anti-fibrinolytic agents, such as tranexamic acid (TA), reduce the risk of death in bleeding trauma patients. On the other hand, it has been suggested that TA administration reduces blood loss and the incidence of postpartum hemorrhage (PPH) in females after vaginal or elective CS verse effects and higher efficacy is needed. Moreover, misoprostol is a prostaglandin E1 analog which has been introduced as a uterotonic agent for preventing PPH following CS. A recent study reported that oral or sublingual misoprostol is more effective than the placebo in reducing severe PPH, following CS

ELIGIBILITY:
Inclusion Criteria:

* women who undergone elective cesarean section (C.S) and exposed to intraoperative bleeding about 500 ml diagnosed by visual analog estimation due to atonic uterus
* age between 18 and 45 years, gestational age of 37-40 weeks, singleton pregnancy, CS with inferior segment incision, and spinal anesthesia.

Exclusion Criteria:

* having an underlying disease (heart, liver, kidney, pulmonary, etc.),
* eclampsia and severe preeclampsia
* allergy to TA (such as known allergy or thromboembolic event during pregnancy) and misoprostol
* coagulation disorders
* refuse or unable to consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women who undergo elective cesarean section (C.S) and exposed to intraoperative bleeding about 500 ml diagnosed by visual analog estimation due to atonic uterus
Enrollment: 150 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
number of patients develop postpartum hemorrhage | 6 hours post operative
  calculation of number of patients develop postpartum hemorrhage

SECONDARY OUTCOMES:
intraoperative blood loss (ml) | during the operation
  calculation of the amount of blood loss in ml by gravimetric methods

OTHER OUTCOMES:
postoperative blood loss (ml) | 6 hours post operative
  calculation of the amount of blood loss in ml by gravimetric methods
number of patients need blood transfusion | 24 hours postoperative
  calculation of number of patients need blood transfusion

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided